CLINICAL TRIAL: NCT00374361
Title: Relationship of Endothelial Function to Insulin Sensitivity in African American and Caucasian Adolescents
Brief Title: Study of the Relationship Between Blood Vessels and Insulin Response in Adolescents
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Ohio State University
Other Study IDs: ENDO 203; AHA 0355195B (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Heart Disease; Stroke
Keywords: insulin sensitivity; endothelial function; adolescence; lipids; puberty
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Heart Diseases; Stroke; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caucasian Adolescents: Caucasian Adolescents
- African-American Adolescents: African-American Adolescents

SUMMARY:
This study is designed to determine whether there is a relationship between the way insulin and blood vessels work. The difference in the interaction between Caucasian and African American adolescents will also be examined. This may play a role in the differing rates of heart disease and diabetes between the two groups.

DETAILED DESCRIPTION:
Purpose: The purpose of the research is to learn more about how the lining of arteries in the body (called the endothelium) and insulin work in adolescents. Abnormalities in how the blood vessels and insulin work in adolescents may cause high blood pressure, type 2 diabetes, stroke and heart disease.

Healthy adolescents between 8 and 18 years of age are being studied in the Ohio State University General Clinical Research Center. Two visits will be necessary. One will be a screening visit to determine the child's stage of puberty and obtain a medical history. The second will be the study visit. During the latter, blood vessel function will be determined by studying the change in forearm blood flow before and after blood flow to the forearm is stopped. Insulin sensitivity will be determined using glucose water given into a vein.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or African American adolescent
* Between 8 and 18 years of age

Exclusion Criteria:

* Pregnancy
* Chronic Disease
* Acute Disease
* Medication Requirement

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents
Sampling Method: Probability Sample
Enrollment: 66
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Hoffman, MD, Study Chair — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Observational

REFERENCES:
- [Result] Hoffman RP. Indices of insulin action calculated from fasting glucose and insulin reflect hepatic, not peripheral, insulin sensitivity in African-American and Caucasian adolescents. Pediatr Diabetes. 2008 Jun;9(3 Pt 2):57-61. doi: 10.1111/j.1399-5448.2007.00350.x. Epub 2008 Jan 21. PMID 18221434
- [Result] Duck MM, Hoffman RP. Impaired endothelial function in healthy African-American adolescents compared with Caucasians. J Pediatr. 2007 Apr;150(4):400-6. doi: 10.1016/j.jpeds.2006.12.034. PMID 17382119
- [Result] Hoffman RP. Increased fasting triglyceride levels are associated with hepatic insulin resistance in Caucasian but not African-American adolescents. Diabetes Care. 2006 Jun;29(6):1402-4. doi: 10.2337/dc06-2460. No abstract available. PMID 16732033
- [Result] Xie L, Hoffman RP, Veng-Pedersen P. Noncompartmental pharmacokinetics analysis of glucose-stimulated insulin response in African-American and Caucasian youths. Biopharm Drug Dispos. 2009 Apr;30(3):117-25. doi: 10.1002/bdd.652. PMID 19288584